CLINICAL TRIAL: NCT00494910
Title: A Randomized Controlled Trial of Group Psychotherapy Interventions for Cancer Patients
Brief Title: Randomized Controlled Trial of Group Psychotherapy Interventions for Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fordham University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-094
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Palliative Care
Keywords: Palliative Care; Terminally Ill; Group Therapy; 07-094

ARMS (2):
- 1 (Experimental): Meaning Centered Group Psychotherapy (MCGP)
  Interventions: Behavioral: Meaning Centered Group Psychotherapy
- 2 (Active Comparator): standardized Supportive Group Psychotherapy
  Interventions: Behavioral: Supportive Group Psychotherapy

INTERVENTIONS:
Behavioral: Meaning Centered Group Psychotherapy — this eight-week (1 ½ hour weekly sessions) Session 1 - Concepts of Meaning and Sources of Meaning Session 2 - Cancer and Meaning Session 3 - Meaning and Historical Context of Life Session 4 - Storytelling, Legacy Project (optional) Session 5 - Limitations and Finiteness of Life Session 6 - Responsibility, Creativity, Deeds Session 7 - Experience, Nature, Art, Humor Session 8 - Transitions, Goodbyes, Hopes for the Future
  Arms: 1
Behavioral: Supportive Group Psychotherapy — The eight weekly 1 ½ hour sessions will focus on group discussion on a set of specific themes that emerge for patients coping with cancer. The session themes or topics will include such issues as: the discussion of strategies for coping with medical issues and procedures, communication with health care providers and issues related to family, friends, and occupational life.
  Arms: 2

SUMMARY:
The purpose of this study is to compare two types of group counseling for cancer patients: Meaning-Centered counseling and Supportive counseling. Many cancer patients seek counseling to help with the emotional burden of their illnesses. Counseling often helps them cope with cancer by giving them a place to express their feelings. "Meaning-Centered" group counseling is intended to teach cancer patients how to maintain or even increase a sense of meaning and purpose in their lives, despite cancer. "Supportive" group counseling is intended to help you cope with cancer by giving you a place to express your feelings and get support from other cancer patients. The purpose of this study is to compare the benefits of these two types of counseling approaches for cancer patients.

DETAILED DESCRIPTION:
To conduct a randomized controlled trial comparing the efficacy of Meaning-Centered Group Psychotherapy (MCGP) versus a standardized Supportive Group Psychotherapy (SGP) in reducing psychological distress (depression and anxiety), end-of-life despair (hopelessness, desire for hastened death, and suicidal ideation), and improving spiritual well-being and overall quality of life in a sample patients with advanced cancer.

To assess the relative impact of Meaning-Centered Group Psychotherapy on different aspects of spiritual well-being (e.g., a sense of meaning and purpose versus spirituality linked to religious faith).

To examine clinical and demographic variables that may correspond to differential responses to Meaning-Centered Group Psychotherapy (e.g., potential mediating and moderating influences such as illness severity, religion and religiosity, level of education, race/ethnicity, level of pre-intervention social support, presence of pain and physical symptom burden).

ELIGIBILITY:
Inclusion Criteria:

* > or = to 21 years of age.
* All patients with stage IV solid tumor cancers; or Stage III solid tumor cancers(excluding breast and prostate cancer) who are receiving ambulatory care at Memorial Sloan-Kettering Cancer Center.
* Able to communicate with an English speaking therapist
* Able to comprehend English to complete study assessments

Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator's judgment, to preclude participation in a group-format intervention (i.e., acute psychiatric symptoms which require individual treatment).
* Presence of cognitive impairment disorder (i.e., delirium or dementia) sufficient, in the investigator's judgment, to preclude meaningful informed consent and/or data collection. The Mini Mental State Examination (MMSE) will be used as a cognitive screening tool. Patients with MMSE scores below 20 will be excluded.
* Karnofsky Performance Rating Scale score below 50 or physical limitations or illness severity sufficient to preclude participation in outpatient group psychotherapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2007-06-26 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
The primary outcomes to be measured include measures of spiritual well-being (meaning) and psychological distress (depression, hopelessness, optimism quality of life). | 16 weeks

SECONDARY OUTCOMES:
To examine clinical and demographic variables that may correspond to differential responses to Meaning-Centered Group Psychotherapy. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Breitbart W, Rosenfeld B, Pessin H, Applebaum A, Kulikowski J, Lichtenthal WG. Meaning-centered group psychotherapy: an effective intervention for improving psychological well-being in patients with advanced cancer. J Clin Oncol. 2015 Mar 1;33(7):749-54. doi: 10.1200/JCO.2014.57.2198. Epub 2015 Feb 2. PMID 25646186
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org